CLINICAL TRIAL: NCT00548106
Title: Evaluation of a New Cow's Milk Infant Formula Containing Partially Hydrolized Whey
Brief Title: Safety Study of Infant Formula With Partially Hydrolized Whey
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn due to the company decision
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Sor461707ctil
Record Dates: First submitted 2007-10-22; First posted 2007-10-23 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2010-07

CONDITIONS: Growth Failure
Keywords: infant formula, milk allergy, hydrolized whey
MeSH Terms: conditions — Failure to Thrive; Milk Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Infants will be fed the new hydrolyzate formula.
  Interventions: Dietary Supplement: partially hydrolyzed whey
- 2 (Placebo Comparator): Nan HA infant formula
  Interventions: Dietary Supplement: partially hydrolyzed whey; Dietary Supplement: Nan HA

INTERVENTIONS:
Dietary Supplement: partially hydrolyzed whey — Total infant feeding by study formula.
  Other Names: Other names are not available yet.
Dietary Supplement: Nan HA — Total infant diet by study formula.
  Other Names: Not available yet.
  Arms: 2

SUMMARY:
The study will be a randomized, double-blind, prospective trial. Newborn infants (enrollment age 0-14 days) will be assigned randomly to receive one of two products, provided in identical packages except for the lid color. Neither the investigators nor the parents will know which product the infant is receiving.

The infants will be monitored at study enrollment, and at 4, 8, and 12 weeks of age.

There will be two study groups, each receiving one of the following formulas:

1. The new partially hydrolyzed whey formula (NF) - Materna cow's milk infant formula containing partially hydrolyzed whey protein, produced and packaged by Materna Laboratories, Maabarot.
2. The currently marketed partially hydrolyzed whey formula (CF) - Nan HA, produced by Nestlé. In order to maintain blinding, the Nan HA will be repacked in packaging identical to the Materna product, except for the lid color

DETAILED DESCRIPTION:
The study will be a randomized, double-blind, prospective trial. Newborn infants (enrollment age 0-14 days) will be assigned randomly to receive one of two products, provided in identical packages except for the lid color. Neither the investigators nor the parents will know which product the infant is receiving.

The infants will be monitored at study enrollment, and at 4, 8, and 12 weeks of age.

There will be two study groups, each receiving one of the following formulas:

1. The new partially hydrolyzed whey formula (NF) - Materna cow's milk infant formula containing partially hydrolyzed whey protein, produced and packaged by Materna Laboratories, Maabarot.
2. The currently marketed partially hydrolyzed whey formula (CF) - Nan HA, produced by Nestlé. In order to maintain blinding, the Nan HA will be repacked in packaging identical to the Materna product, except for the lid color

ELIGIBILITY:
Inclusion Criteria:

Healthy term neonates whose mothers are not able or choose not to breastfeed for medical, social, or personal reasons, will be recruited

Exclusion Criteria:

* Twins
* Premature or low birth weight (< 2500 g).
* Chromosomal abnormalities or congenital malformations.
* Jaundice of more than 12 mg% and/or phototherapy.
* Treatment with antibiotics or other drugs during the last three days or more prior to the commencement of the study.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Growth parameters, colic and bowel movements parameters. | 3 months

SECONDARY OUTCOMES:
Side effects | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Zvi Weizman, MD, Principal Investigator — Head, Pediatric GI and Nutrition Unit
Locations (1):
- Soroka Medical Center, Beersheba, Israel